CLINICAL TRIAL: NCT05873985
Title: The Acute Effect Of Dynamic Taping Applied To The Neck And Back Region On Upper Body Posture In Asymptomatic Male Individuals
Brief Title: The Acute Effect of Dynamic Taping on Upper Body Posture.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Fuat YÜKSEL, Assoc Prof Dr., Gazi University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Efe1
Record Dates: First submitted 2023-05-03; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Dynamic Tape; Postural; Defect

STUDY DESIGN:
Intervention Model Description: double-blind randomized controlled trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic tape on experimental group (Experimental): As a result of randomization, dynamic tape was applied to 25 people with a special technique.
  Interventions: Other: Dynamic tape on experimental group
- Sham tape on placebo group (Placebo Comparator): As a result of randomization, dynamic tape was applied to 26people with a sham technique.
  Interventions: Other: Sham tape on placebo group

INTERVENTIONS:
Other: Dynamic tape on experimental group — The dynamic taping application was carried out in 2 stages. Three "I"-shaped tapes were cut. In the first stage, the person was asked to perform scapular retraction, and in this position, the tape was placed by applying medium tension to the anterior part of the other deltoid muscle, passing from the anterior part of the deltoid muscle to the upper thoracic region. In the second stage, the participant was asked to do scapular retraction and depression, and while maintaining this position, medium tension was applied to the lower thoracic vertebra starting from the anterior part of the deltoid muscle and the acromion and tape was applied. Afterward, this process was applied on the other side
  Arms: Dynamic tape on experimental group
Other: Sham tape on placebo group — Sham taping was performed in 2 stages. Three "I"-shaped tapes were cut. Participants were asked to stand in the comfortable position they used during the day. The first tape was adhered from the starting point of the spine of the scapula with the acromion to the junction of the spine of the scapula and the acromion on the other side without any tension. The other two tapes, starting from the beginning and ending points of the first tape, were adhered to the lower thoracic region without any tension
  Arms: Sham tape on placebo group

SUMMARY:
The aim of this study was to evaluate the acute effect of Dynamic tape on cervical and thoracic region posture in asymptomatic male individuals.

DETAILED DESCRIPTION:
Fifty-one asymptomatic individuals between the ages of 18 and 32 years were included in the study. The participants in this study were randomised into two groups, named "Dynamic Taping" (mean age± sd: 23.28±3.41 yrs, n=25) and "Sham Taping" (mean age± sd: 25.15±4.13 yrs, n=26). In the Dynamic taping group, tapes were applied with optimal stretching, while in the Sham taping group, tapes were applied without any stretch. All measurements were done before taping and 30 minutes after taping. Craniovertebral, cranio-horizontal and sagittal shoulder angles were calculated with photographic posture analysis, while thoracic kyphosis was evaluated with a digital inclinometer (JTech IQ Pro™, ABD).

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18-40 years,
* male gender,
* not having any injuries to the neck and back region in the last 3 months

Exclusion Criteria:

* Individuals who were allergic to taping,
* had neurological or rheumatological disorders
* felt discomfort after starting the study

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Photographic Posture Assessment | 5 minutes before tape
  To take pictures of the participants, the camera (Logitech, Switzerland) was placed on a tripod with a height of 115 cm and at a distance of 1.5 m (33). In order to maintain the same distance between the camera and the participants, a spot on the ground was marked for the subjects to stand, and the tripod was fixed to the ground. The photos were taken of the left side of the subjects in standing position. Before photographing, reflective markers were placed on the lateral canthus, tragus, 7th cervical vertebra, and acromion. During the photography, the subjects were asked to stand in a comfortable position as in daily life.
Photographic Posture Assessment | 15 minutes after tape
  o take pictures of the participants, the camera (Logitech, Switzerland) was placed on a tripod with a height of 115 cm and at a distance of 1.5 m (33). In order to maintain the same distance between the camera and the participants, a spot on the ground was marked for the subjects to stand, and the tripod was fixed to the ground. The photos were taken of the left side of the subjects in standing position. Before photographing, reflective markers were placed on the lateral canthus, tragus, 7th cervical vertebra, and acromion. During the photography, the subjects were asked to stand in a comfortable position as in daily life.
Cranio-horizontal angle (Before) | 5 minutes before tape
  Photographs were analysed using the "ImageJ" program and CH angle were calculated and data were recorded. This procedure was performed by a researcher blinded to the study. This is the angle between the horizontal line drawn from the tragus and the line drawn from the tragus to the lateral canthus of the eye. It provides information about the position of the head above the neck and the location of the upper cervical spine.
Cranio-horizontal angle (after) | 15 minutes after tape
  Photographs were analysed using the "ImageJ" program and CH angle were calculated and data were recorded. This procedure was performed by a researcher blinded to the study. This is the angle between the horizontal line drawn from the tragus and the line drawn from the tragus to the lateral canthus of the eye. It provides information about the position of the head above the neck and the location of the upper cervical spine.
Craniovertebral angle (before) | 5 minutes before tape
  Photographs were analysed using the "ImageJ" program and CV angle were calculated and data were recorded. This procedure was performed by a researcher blinded to the study.This is the angle between the horizontal line drawn from the 7th cervical vertebra and the line drawn from the 7th cervical vertebra to the tragus . The CV angle provides information about the position of the lower cervical region and is used in the objective evaluation of FHP.
Craniovertebral angle (after) | 15 minutes after tape
  Photographs were analysed using the "ImageJ" program and CV angle were calculated and data were recorded. This procedure was performed by a researcher blinded to the study.This is the angle between the horizontal line drawn from the 7th cervical vertebra and the line drawn from the 7th cervical vertebra to the tragus . The CV angle provides information about the position of the lower cervical region and is used in the objective evaluation of FHP.
Sagittal shoulder posture angle ( Before) | 5 minutes before tape
  Photographs were analysed using the "ImageJ" program and SSP angle were calculated and data were recorded. This procedure was performed by a researcher blinded to the study.This is the angle between the horizontal line drawn from the acromion and the line connecting the acromion to the 7th cervical vertebra. This assessment provides information about the position of the shoulder
Sagittal shoulder posture angle (after) | 15 minutes after tape
  Photographs were analysed using the "ImageJ" program and SSP angle were calculated and data were recorded. This procedure was performed by a researcher blinded to the study.This is the angle between the horizontal line drawn from the acromion and the line connecting the acromion to the 7th cervical vertebra. This assessment provides information about the position of the shoulder

SECONDARY OUTCOMES:
Thoracic kyphosis angle (Before) | 5 minutes before tape
  TK angle was measured with a dual digital inclinometer (JTech IQ Pro™, USA). Participants were asked to stand in a relaxed position. The dual inclinometer device was placed over the spinous processes of the 1st thoracic vertebra and the 12th thoracic vertebra. The measured angle was recorded as the TK angle.
Thoracic kyphosis angle (after) | 15 minutes after tape
  TK angle was measured with a dual digital inclinometer (JTech IQ Pro™, USA). Participants were asked to stand in a relaxed position. The dual inclinometer device was placed over the spinous processes of the 1st thoracic vertebra and the 12th thoracic vertebra. The measured angle was recorded as the TK angle.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No